CLINICAL TRIAL: NCT07149610
Title: Connected Care for Type 2 Diabetes: a Study Protocol for a Structured Self-Management Intervention Through Technology and Healthcare Collaboration
Brief Title: Connected Care for Type 2 Diabetes Self-Management
Acronym: RCT_SM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marche Region Regional Health Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4197
Record Dates: First submitted 2025-08-07; First posted 2025-09-02 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Type 2
Keywords: self-management; digital solution; Diabete type 2; Chronic diseases; glycated hemoglobin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease

STUDY DESIGN:
Intervention Model Description: A multicentric, open-label, two-arms randomized controlled trial (RCT) will be conducted to evaluate the improvement of self-management abilities of patients affected by T2DM, after the implementation of the m-health solution (medical device) (treated group), versus usual care (control group). The outcomes assessments will be carried at baseline and at 6, 12 and 18 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group (utilizing m-health solution) (Active Comparator): The participants assigned to the treated group, in addition to the regular T2DM care, will be provided with a m-health solution to support the SM of T2DM, aimed to improve their SM' skills and abilities. The m-health solution will allow the patients to:
  1. track their data, such as glycaemic status, blood pressure, therapy, steps and physical activity, sleep, body weight, laboratory tests (HbA1c, creatinine, cholesterol, etc.);
  2. check the target values defined by the diabetologist (e.g., blood glucose, HbA1c, lipid profile, etc.);
  3. view their treatment plan;
  4. view the diet indicated by the dietitian and record meals/calculate calories/carbohydrates in a simple way (e.g., through list of foods with pictures of dishes and portions);
  3) receive alerts (e.g., therapy reminders) and motivational messages; 4) view summary statistics; 5) communicate with the HCPs through a chat; 6) fill out surveys; 7) access to educational material and technical assistance;
  Interventions: Device: M-health solution classified as Class I Medical Devices, equipped with a CE certificate. The m-health solution will be integrated with the EPR currently used by the CADs of the Marche region
- Control group (attending usual T2DM care) (No Intervention): The patients assigned to the control group will receive regular T2DM care according to the Diabetes Association standards

INTERVENTIONS:
Device: M-health solution classified as Class I Medical Devices, equipped with a CE certificate. The m-health solution will be integrated with the EPR currently used by the CADs of the Marche region — The m-health solution used in the study includes the following interfaces:
  1. for the HCPs of the CADs:
     * a section of the EPR currently used (Metaclinic), to set the mobile application and to collect clinical data recorded by the patients;
     * a software to develop and monitor personalised diets (MetaDieta);
  2. for the patients: two mobile applications, one for the monitoring of the clinical data and life style (DiaWatch Meteda) and one for the monitoring of the diet (MyDiet), with the latter accessible from a 'button' included in the first one.
  The HCPs of the CADs, already having access to the EPR Metaclinic, will access a dedicated section for the setting of the target values and goals (e.g., glycaemia, physical activity, etc.) and for the activation of the app DiaWatch Meteda. After the connection of the app with Metaclinic, the data registered in the apps by the patients will be visible by the HCPs in the EPR dashboard.
  Arms: Treated group (utilizing m-health solution)

SUMMARY:
The primary objective of this Randomized Clinical Trial is to improve the self-management (SM) competencies of patients affected by Type 2 Diabetes Mellitus (T2DM) living in the Marche region (Italy) through the support of a mobile health (m-health) solution personalised by the diabetologist and integrated with the Electronic Patient Record (EPR), assessed through the change in glycated haemoglobin (HbA1c) levels (%) from baseline to the end of the intervention (primary outcome).

Researchers will compare the use of the m-health solution (treated group) to usual T2DM care (control group) in determining change in HbA1c levels (%). The intervention will start at the Diabetic Centres (CADs) where patients are currently followed up and will then take place in each participant's home

Participants of the treated group will:

* receive dedicated training on the use of the m-health solution
* receive the personalization of the m-health solution
* use the m-health solution to: 1) track and view the data related to their health status (e.g., glycaemic status, lifestyle habits, diet) and treatment plane; 2) receive alerts and motivational messages; communicate with the Health Care Professionals (HCPs) of the Diabetic Centre (CAD) in case of need; 3) access to the educational material and to the technical assistance, when needed.

HCPs will be able to monitor the patients' data and clinical parameters and to communicate with the patients. After a baseline evaluation (T0), three follow-up evaluations will be conducted at 6, 12 and 18 months (T1-T2-T3 respectively) , during the usual physician' visits, as part of clinical routine.

The evaluation phases (T0, T1, T2, T3) will be conducted through data derived from: 1) self-administered and paper-based questionnaires, validated in the Italian language; 2) the clinical assessment of patients; 3) the m-health solution, as data automatically derived from the m-health solution; 4) a focus group carried out in a subsample of participants.

Data regarding different health-related areas (T2DM severity; medication adherence; lifestyle habits; self-efficacy related to management of the disease; quality of life), usability of the m-health solution, participants' experience with the intervention, utilization of the m-health solution by the patients, and the cost-effectiveness of the intervention, will be evaluated.

Patients participating in the study will not be required to make any additional visits or undergo any laboratory analysis beyond those specified in their therapeutic plan.

DETAILED DESCRIPTION:
1. Details about recruitment: Prior to the start of the study, the medical directors, the nursing healthcare managers, and nursing coordinators of the CADs involved in the study will be informed about characteristics, methods and aims of the research. The principal investigator (PI) of the study will be responsible to conduct a specific training session on the protocol, the procedures and the data collection to all the HCPs of the CADs participating in the study as staff (e.g., doctors, dietician, nurses), to ensure standardised procedures across all the participating centres and without interfering with clinical-assistance and other priority activities. At the same time, the owners of the mhealth solution will provide specific training on the use of m-health solution, including the interface integrated with the EPR and the mobile app for the patients. In details, the company contact person, in collaboration with the scientific coordinator of the company, will held an in-presence training session of 1 hour for the HCPs, in a dedicated time before the start of the study, to be conducted in small groups, in an interactive way, accepting and answering any doubts. This educational session will include a theorical component, regarding characteristics, functionalities and potentialities of the m-health solution, and a practical component, based on simulations about the use of the m-health solution and about an example of training that will be provided to the participants. The necessity to strengthen and/or supplement the training will be evaluated by the owners of the m-health solution, and, eventually, faced.

The information letter and the paper-based consent form will be delivered by the investigators to the eligible patients, in the CADs of the Marche Region involved in the study, making themselves available for clarifications and explanations. The participants will be enrolled only after having been deeply informed about modalities and principles of data treatment, along with the aims and the characteristics of the study, and only after signing the paper-based informed consent form for the authorization of data processing and for voluntary participation in the study, after a reflection period of 2 weeks. The participants having signed the informed consent to participate in the research will be invited by the investigators, through telephonic calls and/or emails, to consult one of the diabetologist participating as staff in the study. The doctors will carry out the visits to attest the eligibility of the participant for the study, with the support of other HCPs of the CADs, such as nurses, based on the inclusion criteria. The doctor will sign the consent forms too, making him-/her-self available to provide further details and to solve any doubts of the patients. Each signature will be personally dated by each signatory, and the informed consent and any additional patient information will be retained by the investigator. A signed copy of the informed consent and information sheet will be given to each patient. Participants who have signed the consent form but whose inclusion criteria are not confirmed by the doctor will not be included in the study.

2- Legal, ethical and technical considerations:

This study, and, consequently, the data collection, usage and storage procedures, will be conducted according to the principles expressed in:

* The Declaration of Helsinki 2024
* the standards of Good Clinical Practice
* the Legislative Decree no. 196/03 Italian Personal Data Protection Code
* EU General Data Protection Regulation 2016
* Legislative Decree No. 101/2018 on Provisions for the adaptation of national legislation to the provisions of European Regulation 2016/679
* Guidelines for the collection of informed consent for participation in clinical trials, National Coordination Centre for Ethics Committees.

The study will start only after notification and acknowledgement by the Regional Ethics Committee and the completion of the administrative requirements of the institution where the study is being conducted. No sponsorship is envisaged for the conduction of this study

ELIGIBILITY:
Inclusion Criteria:

* patients with T2DM (as confirmed by the physician's diagnosis);
* belonging to one of the 13 Diabetes Centres (CADs) of the Marche region in Italy (Pesaro, Urbino, Fano, Senigallia, Jesi, Fabriano, IRCCS-INRCA, Azienda Ospedaliera Universitaria delle Marche, Civitanova Marche, Macerata, Fermo, San Benedetto del Tronto e Ascoli Piceno);
* age > = 18;
* resident in the Marche region;
* HbA1c > 7 on most recent laboratory report within the last 3 months;
* no changes in diabetes medication in the previous 6 months;
* no prescription for any hypoglycaemic agent within the previous 4 weeks or taking a consistent dose of one or more oral hypoglycaemic agents for more than 12 weeks;
* owning smartphone/mobile phone with an internet connection;
* capable to consent;
* fulfilling and signing the informed consent;
* with self-reported competencies of communicating verbally in local language (corresponding to a level of Italian language knowledge =>A2 of the CEFR levels).

Exclusion Criteria:

* acute medical problems: myocardial infarction or stroke within 6 months, difficulty in exercise and physical activity due to spinal disease (intervertebral disc prolapse, spinal stenosis, etc.), joint disease, or major surgery at the time of screening, painful arthritis, spinal stenosis, amputation, painful foot lesions or neuropathy limiting balance and mobility, advanced Parkinson's disease and/or neuromuscular disorders, advanced dementia, metastatic cancer, in long-term immunosuppressant therapy, significant visual or hearing impairment, uncontrolled hypertension or other serious conditions that restrict their participation in the study, severe/major depression and other relevant psychiatric disorders;
* estimated glomerular filtration rate < 30 mL/min/1.73 m2;
* plan to receive surgery that could limit physical activity during the study period;
* pregnant or breastfeeding;
* participation in another studies;
* lack of written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To improve the SM competencies of patients affected by T2DM living in the Marche region through the support of a m-health solution personalized by the diabetologist and integrated with the EPR of patients. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through the change in HbA1c levels (%)

SECONDARY OUTCOMES:
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed evaluating the change in the level of fasting glucose (mg/dl)
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed evaluating the change in glycaemic variability/capillary blood glucose monitoring, when foreseen by patients' therapeutic plan
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed evaluating the change in the levels of Serum total cholesterol (mg/dl), triglycerides (mg/dl), High-Density Lipoproteins (mg/dl) and Low-Density Lipoproteins cholesterol (mg/dl).
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 12 and at month 18.
  This outcome will be assessed evaluating the change in Microalbuminuria levels (mg/dl).
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed evaluating the change in waist circumference (cm)
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through evaluating the body weight (kg).
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed evaluating the change Body Mass Index (BMI) (kg/m^2).
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed evaluating the change in blood pressure's values (mmHg);
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed evaluating changes regarding the following anamnestic measurements: comorbidities, medications and complications related to T2DM, including the number of hypoglycaemia and hyperglycaemia episodes in the last 6 months.
To evaluate the changes, after the intervention, in T2DM severity, through clinical records/physician visits. | This outcome will be evaluated from HADs, at baseline (month 0) and at the the end of treatment (namely at month 18).
  This outcome will be assessed evaluating the number of unscheduled hospital visits due to hypoglycaemia or hyperglycaemia within 12 months: outcome assessed retrospectively through the Administrative Healthcare Databases (HADs) of Hospital discharge records occurred in public and private hospitals and Emergency and Urgency care according to ICD-9 codes (250.3, 250.8, 251.0, 251.1, 251.2, 270.3, 790.6).
To evaluate the changes, after the intervention, in the levels of medication adherence | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through the "Medication Adherence Report Scale- MARS-5 ©", validated in Italy, composed by five questions on both unintentional and intentional non-adherence, namely forgetting, changing dosage, stopping, skipping and taking less medication. The score ranges from 5 to 25, where a higher score indicates higher self-reported adherence.
To evaluate the changes, after the intervention, in dietary and alcohol consumption habits | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through the questionnaire "Literature Based Adherence Score to Mediterranean Diet- MEDILITE", that enables the user to ascertain their consumption of 9 food categories, defined in scientific studies examining the correlation between adherence to the Mediterranean diet and health outcomes. The 9 food groups are: fruits; vegetables; cereals; legumes; fish; meat and meat products; dairy products; alcohol; olive oil. The scores assigned differ for each item: typical foods of the Mediterranean diet (2=highest consumption category; 1=intermediate category; 0=lowest category); non-typical foods (2=lowest intake; 1=intermediate intake; 0=highest consumption); alcohol (2=1-2 alcohol units/day; 1=1 alcohol unit/day; 0= >2 alcohol units/day); olive oil (2=regular use; 1=frequent use; 0=occasional use). The final score, obtained from the sum of all these scores, ranges from 0 (low adherence to the Mediterranean diet) to 18 (high adherence).
To evaluate the changes, after the intervention, in smoking habits | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through n. 11 ad hoc questions to analyse the smoking habits and history, elaborated from the questions included in the EPR of patients (routinely collected) and from the National Institute of Statistics-ISTAT questionnaires.
To evaluate the changes, after the intervention, in levels of physical activity | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through the "International Physical Activity Questionnaire- Short Form- IPAQ-SF": validated in Italian language, evaluates frequency (days per week) and duration (minutes per day) of three types of activity, i.e., walking, moderate intensity and vigorous intensity activities. The scale assigns a score to each activity and a total score, calculated from the duration and frequency of three activities. Activity volume can also be expressed in MET-minutes (METs x minutes x frequency per week). Scores can be continuous or categorized:
  1. Low - below moderate or high criteria;
  2. Moderate - e.g., 3+ days of vigorous activity (20+ min/day), or 5+ days of moderate/walking (30+ min/day), or 600+ MET-min/week;
  3. High - 3+ days vigorous activity totaling 1500+ MET-min/week, or 7+ days of mixed activity reaching 3000+ MET-min/week.
To evaluate the changes, after the intervention, in the levels of self-efficacy perceived by partecipants | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through the "The Italian Diabetes Management Self-Efficacy Scale- IT-DMSES", that consists of 15 items divided into two factors of self-efficacy in diabetes management: 1) self-perception of patient's ability to manage the activities related to diabetes management (e.g., medication adherence, Glycaemic Control), and 2) self-efficacy in lifestyle management (e.g., eating behaviours, physical activities). Scores per factor range from 0 to 10, indicating low (0-3), mid (4-6), and high (7-10) levels of self-efficacy.
To evaluate the changes, after the intervention, in the levels of quality of life perceived by partecipants | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through the scale "EuroQol 5-digit 5-level Visual Analogue Scale- EQ-5D-5L VAS", validated in Italian language, in details through its descriptive system, consisting on five dimensions: mobility, independence, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no/mild/moderate/severe/extreme problems. The participant is asked to indicate his/her health status with the most appropriate statement in each of the five dimensions, producing also a 5-digit number that describes the health profile of the participant.
To evaluate the changes, after the intervention, in the levels of quality of life perceived by partecipants | This outcome will be evaluated from baseline to the end of treatment, in details, at month 0, at month 6, at month 12 and at month 18.
  This outcome will be assessed through the scale "EuroQol 5-digit 5-level Visual Analogue Scale- EQ-5D-5L VAS", validated in Italian language, in details through the EQ VAS part, represented in a vertical scale from 0 to 100 in 5-point increments. The participant is asked to represent his/her health status putting a cross on the scale, then translated into an integer between 0 and 100.
To collect information regarding participants' perception of usability of the m-health solution, their level of satisfaction and any benefits they have experienced. | This outcome will be evaluated at month 6, at month 12 and at the end of the intervention (namely at month 18).
  This outcome will be through the Italian version of the System Usability Scale-SUS" , a ten-item tool giving a global view of subjective assessments of usability. The response options are based on the Likert scale, from 1= strong disagreement; to 5= strong agreement, for a total score ranging from 0 to 100, to be evaluated based on a computation table.
To collect information regarding participants' experience with the intervention. | This outcome will be evaluated at the end of the intervention, namely at month 18
  This outcome will be assessed through focus groupm carried out in a subsample of participants (max 5-10 participants for each focus group) to gain additional insights on the patient's experience with the intervention, that will allow patients to discuss about perceptions and opinions about the utility of the intervention and of the m-health solution, letting patients free to express their ideas and suggestions. The focus group will be carried out by two experienced researchers from the research team: 1) the moderator, acting as initiator and facilitator of the discussion, as well as mediating between participants and conducting discussion through posing main questions; 2) the observer/note-taker, acting as rapporteur, writing down notes about both discussion between participants (e.g., topics covered, opinions emerging, contrasts, new issues). The discussion will be audio recorded and transcribed verbatim to facilitate subsequent analysis and reporting.
To collect information regarding the utilization of the m-health solution by the patients | This outcome will be evaluated at month 6, at month 12 and at the end of treatment, namely at month18
  This outcome will assessed through data analytics collected by the digital system as utilization measures automatically derived from the mobile apps used by the patients, namely, number of accesses, time of use, and frequency of use of the key features such as inputs of data, access to training/information documents, chat, and consultation of target values and treatment plan.
  The data collected will be processed to produce periodic reports highlighting areas of increased use, any critical issues, and suggestions for future improvements.
To evaluate the cost-effectiveness of the intervention. | This outcome will be evaluated at the end of the intervention, namely at 18 months
  This outcome will be assessed through Incremental Cost-Effectiveness Ratio (ICER), that will be calculated as the difference in costs divided by the difference in health benefits over an 18-month period from a healthcare sector perspective. A bottom-up micro-costing approach will assess all individual-level costs for control and intervention groups, including diabetes care (hospital admissions, emergency care, outpatient visits, lab tests, drugs, consumables). The intervention group also includes technology-related costs (software, maintenance). The evaluation is within-trial. Cost-effectiveness is based on HbA1c; QALYs, derived from EQ-5D-5L, are used for cost-utility analysis. ICERs will be reported with 95% confidence intervals via bootstrapping. A €25,000-€60,000 per QALY threshold and sensitivity analyses with acceptability curves will assess uncertainty.

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - Diabetic Center of Azienda Ospedaliero Universitaria delle Marche, Ancona, Ancona
  - Diabetic Center of National Institute for the Care and Treatment of the Elderly (Istituto Nazionale di Ricovero e Cura per Anziani-INRCA), Ancona, Ancona
  - Diabetic Center of Territorial Healthcare Authority of Ancona province, Fabriano, Ancona
  - Diabetic Center of Territorial Healthcare Authority of Ancona province, Iesi, Ancona
  - Diabetic Center of Territorial Healthcare Authority of Ancona province, Senigallia, Ancona
  - Diabetic Center of Territorial Healthcare Authority of Ascoli Piceno province, Ascoli Piceno, Ascoli Piceno
  - Diabetic Center of Territorial Healthcare Authority of Ascoli Piceno province, San Benedetto del Tronto, Ascoli Piceno
  - Diabetic Center of Territorial Healthcare Authority of Fermo province, Fermo, Fermo
  - Diabetic Center of Territorial Healthcare Authority of Macerata province, Civitanova Marche, Macerata
  - Diabetic Center of Territorial Healthcare Authority of Macerata province, Macerata, Macerata
  - Diabetic Center of Territorial Healthcare Authority of Pesaro Urbino province, Fano, Pesaro-Urbino
  - Diabetic Center of Territorial Healthcare Authority of Pesaro Urbino province, Pesaro, Pesaro-urbino
  - Diabetic Center of Territorial Healthcare Authority of Pesaro Urbino province, Urbino, Pesaro-Urbino

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP